CLINICAL TRIAL: NCT03540485
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of Melatonin Administration in Patients with Multiple Progressive Primary Sclerosis
Brief Title: Safety and Efficacy of Melatonin in Patients with Multiple Progressive Primary Sclerosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MELATOMS-1; 2018-001779-18 (EudraCT Number)
Record Dates: First submitted 2018-05-04; First posted 2018-05-30 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Sclerosis, Multiple; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Autoimmune Diseases
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Autoimmune Diseases | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): Daily administration of 100 mg of melatonin orally, for 24 months, single dose of melatonin between 10pm to 11pm
  Interventions: Drug: Melatonin
- Control (Placebo Comparator): Daily administration of placebo orally, for 24 months between 10pm to 11pm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin — Daily administration of 100 mg of melatonin orally, for 24 months, single dose of melatonin between 10pm to 11pm
  Arms: Melatonin
Other: Placebo — Daily administration of placebo orally, for 24 months between 10pm to 11pm
  Arms: Control

SUMMARY:
Phase I / II randomized, double-blind, placebo-controlled clinical trial to evaluate the safety and efficacy of melatonin administration combined with ocrelizumab in patients with Progressive Multiple Primary Sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis (MS), the most common inflammatory disease of the central nervous system in young adults, has a huge social and health interest, especially the primary progressive (PP-) course, in which the disability is very fast accumulated and currently there are no available treatments in Spain. PP-MS is characterized by neuro-inflammation and, especially, by neurodegeneration, with brain atrophy as key feature. It has been proposed that PP-MS therapies should combine anti-inflammatory and neuroprotective activities. The investigators have shown that melatonin, an immunomodulatory, antioxidant and neuroprotective compound, ameliorates the disease and modulates the pathogenic/protective immune responses in a MS animal model. Moreover, melatonin caused a long-term improvement of disability on a PP-MS patient. Thus, melatonin could be of interest in the therapy of PP-MS.

So far, ocrelizumab, recently authorized by the European Medicines Agency and incorporated into the portfolio of the Spanish National Health System in December 2018, is the only therapy that has shown some therapeutic efficacy on the decrease in long-term disability.

The purpose of this study is to determine the feasibility of using melatonin combined with ocrelizumab to treat PP-MS. Thus, the investigators propose a randomized, single-blind, placebo-controlled study on the safety and efficacy of melatonin combined with ocrelizumab on PP-MS patients. The investigators will assess the daily administration to patients treated with ocrelizumab for at least 9 months of one oral dose of melatonin containing 100mg during 24 months on patients safety and its effects over brain atrophy progression, Expanded Disability Status Scale scores, quality of life, MS symptoms, circadian impairment and levels of markers of central nervous system inflammation, axonal damage, Blood-brain barrier disruption and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

Patients who come to the Multiple Sclerosis Unit of the Department of Neurology of the Virgen Macarena University Hospital (Seville) or Vithas Nisa Seville Hospital or Virgen del Rocío University Hospital (Seville), and who meet the following criteria:

* Have progressive primary multiple sclerosis according to McDonald's diagnostic criteria modified in 2010.
* Age between 18 and 65 years old.
* Neurological impairment measured with the Expanded Disability Status Scale (EDSS) scale between 2 and 7 (both included, without disability or only clinical symptoms up to ambulatory capacity with bilateral support).
* Not having received any immunomodulatory, except for ocrelizumab in stable doses for at least 9 months before inclusion in this study, or immunosuppressive treatment (including cytostatic agents) during the 3 months prior to participation in the trial.
* If there is a possibility of pregnancy (in women of childbearing age (15 to 44 years)) or paternity, accept the use of a highly effective method of birth control recommended by the Clinical Trial Facilitation Group (CTFG) during the treatment phase of the trial..
* Not having consumed melatonin or other dietary supplements (antioxidants or vitamins (tripling the recommended daily doses) during the month prior to participation in the trial.
* Ability to give informed consent and comply with the visits scheduled in the study.

Exclusion Criteria:

* Alternative diagnosis that explains both the neurological disability and the findings in nuclear magnetic resonance.
* Clinically significant medical problems that, in the opinion of the investigators, may cause tissue damage in the central nervous system or limit its repair, or that may expose the patient to unjustified risks or damages, or cause the patient not to complete the study.
* Clinical history of hypersensitivity reactions to melatonin.
* Pregnancy or lactation, or planning to become pregnant or patients of childbearing age not subject to birth control methods (recommended by the Clinical Trial Facilitation Group (CTFG)).
* Abnormal results in basal blood tests, defined as:
* Serum levels of alanine transaminase or aspartate transaminase greater than 1.5 times the upper limit of normal values.
* Total leukocyte count less than 3,000 / mm3.
* Platelet count less than 85,000 / mm3.
* Serum creatinine level greater than 2.0 mg / dL or glomerular filtration rate less than 30.
* Neurological deterioration measured with the Expanded Disability Status Scale scale of less than 2 or greater than 7.
* Be receiving any immunosuppressive therapy, except for ocrelizumab, including cytostatic agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rates of neurological impairment | 2 years
  Individualized rates of disease progression will be quantified using the rates of neurological impairment (Kurtzke Expanded Disability Status Scale). The scale provides a total score on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability.
Rates of disability | 2 years
  Individualized rates of disease progression will be also quantified using the rates of disability (Multiple Sclerosis Functional Composite - MSFC scale).The MSFC measures are administered in person by a trained examiner. The MSFC can produce scores for each of the three individual measures (measure leg function/ambulation, arm/hand function, and cognitive function) as well as a composite score. Total administration time for all three measures should be approximately 20-30 minutes. Scores on component measures are converted to standard scores (z-scores), which are averaged to form a single MSFC score.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | monthly from date of randomization until the end of the follow-up, assessed up to 24 months
  To determine the incidence of adverse events and any abnormal laboratory values
Cerebral atrophy | In every study visit, assessed up to 24 months
  Cerebral atrophy will be measured through magnetic resonance imaging
Fatigue | In every study visit, assessed up to 24 months
  Fatigue will be assessed using the Modified Fatigue Impact Scale scale (MFIS), a modified form of the Fatigue Impact Scale (Fisk et al, 1994b) based on items derived from interviews with multiple sclerosis patients concerning how fatigue impacts their lives. The total score for the MFIS is the sum of the scores for the 21 items. Items on the MFIS can be aggregated into three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities.
Quality of life using the Multiple Sclerosis International Quality of Life scale | In every study visit, assessed up to 24 months
  Quality of life will be assessed using the Multiple Sclerosis International Quality of Life (MusiQoL) scale, a self-administered and multidimensional questionnaire designed to reflect the point of view held by patients with MS on how the disease affects their daily life. Questionnaire comprises 31 items describing nine dimensions: Activities of Daily Living, Psychological Well-Being, Symptoms, Relationships with Friends-Family-Healthcare System, Sentimental and Sexual Life, Coping and Rejection. Each item was scored on a six-point Likert scale: score of 1 (never ⁄not at all), 2 (rarely ⁄a little), 3 (sometimes ⁄somewhat), 4 (often ⁄ a lot), 5 (always ⁄ very much) and 6 (not applicable).
Sleep disorders | In every study visit, assessed up to 24 months
  The assessment of sleep disorders will be conducted through the Pittsburgh Sleep Quality Index.
Spasticity | In every study visit, assessed up to 24 months
  Spasticity will be analyzed using the Ashworth scale that tests resistance to passive movement about a joint with varying degrees of velocity.
  Scores range from 0-4, with 5 choices. A score of 1 indicates no resistance, and 5 indicates rigidity.
  0 (0) - No increase in tone
  1. (1) - Slight increase in tone giving a catch when the limb was moved in flexion or extension
  2. (2) - More marked increase in tone but limb easily flexed
  3. (3) - Considerable increase in tone - passive movement difficult
  4. (4) - Limb rigid in flexion or extension.

OTHER OUTCOMES:
Efficacy of neuroinflammation | Day 0 and after 2 years
  Neuroinflammation marker CXCL13 will be measured through the human CXCL13 / BLC / BCA-1 Quantikine ELISA Kit (R & D Systems).
Axonal damage | Day 0 and after 2 years
  The levels of the axonal damage marker Neurofilament of the light chain (NfL) will be measured by the NF-light ELISA (UmanDiagnostics).
Oxidative stress | Day 0 and after 2 years
  Oxidative stress will be quantified through the analysis of the total antioxidant capacity (TAC) that will be evaluated through the OxiSelect Total Antioxidant Capacity (TAC) Assay Kit (CellBiolabs, Inc.).
Impact on microbiota | 2 years
  Comparison of biological alpha and beta diversity of the intestinal microbiota of both study groups (classical and optimized antibiotherapy). Calculation of alpha diversity (OTUs richness and Shannon diversity indexes observed, Faith's Phylogenetic Diversity and Evenness) and beta diversity (Jaccard distance, Bray- Curtis distance, Unweighted UniFra distance, used for comparing biological communities) indexes by QIIME 2 (microbiome bioinformatics platform).

CONTACTS AND LOCATIONS:
Overall Officials: Clara M Rosso Fernández, MD/PhD, Principal Investigator — Clinical Research and Clinical Trials Unit (Virgen del Rocío University Hospital, Seville); Antonio Carrillo Vico, PhD, Study Director — Institute of Biomedicine of Seville (IBiS)
Locations (3):
- Spain (3):
  - Virgen Macarena Hospital, Seville, Seville
  - Virgen del Rocio University Hospital, Seville, Seville
  - Hospital Vithas Nisa Sevilla, Seville, Seville

IPD SHARING:
Plan to Share IPD: No